CLINICAL TRIAL: NCT00717392
Title: Evaluation of the Efficacy of Hippotherapy for Children With Developmental Disorders
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Lidia Gabis MD, Director, The Weinberg Child Development Center, Sheba Medical Center
Other Study IDs: SHEBA-08-5327-LG-CTIL
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder
Keywords: ADHD; ASD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Hippotherapy_ADHD: 10 children with ADHD who receive hippotherapy
- Hippotherapy_ASD: 10 children with ASD who receive hippotherapy
- Control_ADHD: 10 children with ADHD who DO NOT receive hippotherapy
- Control_ASD: 10 children with ASD who DO NOT receive hippotherapy

SUMMARY:
Hippotherapy is every program of horseback riding meant to treat people with physiological, mental, social, cognitive or behavioral problems. The purpose of the current research is to evaluate the efficacy of hippotherapy for children with developmental disabilities. The hypothesis is that children with developmental disabilities who are treated with hippotherapy will show better outcomes than children with the same problems who are not treated with hippotherapy.

DETAILED DESCRIPTION:
Hippotherapy is every program of horseback riding meant to treat people with physiological, mental, social, cognitive or behavioral problems. Most studies that tested hippotherapy were uncontrolled and focused on motor problems, such as cerebral palsy. Today, hippotherapy is used for various developmental problems such as Attention deficit / Hyperactivity disorder (ADHD) and Autism spectrum disorder (ASD), without clear information about its efficacy for these populations.

The purpose of the current research is to evaluate the efficacy of 6 months of hippotherapy for children with developmental disabilities. The hypothesis is that children with developmental disabilities who are treated with hippotherapy for 6 months will show better outcomes than children with the same problems who are not treated with hippotherapy.

Assessment:

* BRIEF questionnaire
* Stony Brook Questionnaire

All questionnaires will be applied at the beginning of the study and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age: 5-17 years.
* A diagnosis of ADHD or ASD.

Exclusion Criteria:

* None.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hippotherapy subjects will be taken from horseback riding farms. Control subjects will be taken from a tertiary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Improving the parameters of autism | Repetitive behaviors
  Repetitive behaviors Eye contact Communication

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Gabis, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Weinberg Child Development Center, Sheba Medical Center, Tel-Hashomer, Ramat Gan, Israel